CLINICAL TRIAL: NCT06971536
Title: A Human Clinical Trial on the Pharmacokinetics and Safety of Oral Micellar Green Tea Extract
Brief Title: Safety and Bioavailability of Micellar Green Tea Extract
Acronym: GT Safety & BA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-11-002GT
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Bioavailability and Pharmacokinetics; Safety
Keywords: pharmacokinetics; green tea extract; bioavailability; safety; micellar delivery system

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to interventions in a crossover design to assess the pharmacokinetics over 48 hours; subsequently, the safety of LipoMicel Green tea intervention with the higher bioavailability is evaluated in a subsequent single-arm, 30-day trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Green Tea (Experimental): Each participant receives their treatment i.e., Standard Green Tea hard gel capsules at a total dose of 300 mg green tea extract. Treatments are consumed with a glass of water (approx. 200mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 48 hours post-dose. A washout period of at least 7 days between each treatment is used.
  Interventions: Dietary Supplement: Standard Green Tea
- Phytosome Green Tea (Experimental): Each participant receives their treatment i.e., Phytosome green tea hard gel capsules at a total dose of 250 mg green tea extract. Treatments are consumed with a glass of water (approx. 200mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 48 hours post-dose. A washout period of at least 7 days between each treatment is used.
  Interventions: Dietary Supplement: Phytosome Green Tea
- LipoMicel Green Tea (Experimental): Each participant receives their treatment i.e., LipoMicel green tea soft gel capsules at a total dose of 300 mg green tea extract. Treatments are consumed with a glass of water (approx. 200mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at different time points up to 48 hours post-dose. A washout period of at least 7 days between each treatment is used.
  Interventions: Dietary Supplement: LipoMicel Green Tea

INTERVENTIONS:
Dietary Supplement: Standard Green Tea — A maximum single dose of 300 mg green tea (hard gel capsules)
  Arms: Standard Green Tea
Dietary Supplement: Phytosome Green Tea — A maximum single dose of 250 mg green tea (hard gel capsules)
  Arms: Phytosome Green Tea
Dietary Supplement: LipoMicel Green Tea — A maximum single dose of 300 mg green tea (soft gel capsules)
  Arms: LipoMicel Green Tea

SUMMARY:
This study seeks to determine the short-term effects of daily oral supplementation of LipoMicel Green Tea on oral absorption and safety of green tea in healthy volunteers.

The primary objective is to evaluate and compare the pharmacokinetics of LipoMicel Green Tea (LGT) with that of a standard green tea extract formulation as well as a phytosomal green tea formulation. The secondary objective is to evaluate the safety of LGT in healthy human participants over a 30-day study period.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 21-65 years
* healthy, good physical condition
* voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* use of anti-inflammatory or non-steroidal anti-inflammatory drugs
* previous history of cardiovascular disease or acute or chronic inflammatory disease
* use of antioxidant supplements or cholesterol-lowering agents
* change of diet habits or lifestyle (diet, physical activity, etc.)
* alcohol or substance abuse history
* use of nicotine or tobacco
* participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24, 48 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested green tea extract in healthy adult volunteers and compare the Area under the plasma concentration versus time curve (AUC) with that of other capsules containing green tea extract.
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24, 48 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested green tea extract in healthy adult volunteers and compare the peak plasma concentration (Cmax) with that of other capsules containing green tea extract.
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 12, 24, 48 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested green tea extract in healthy adult volunteers and compare the time point of maximum plasma concentration (Tmax) with that of other capsules containing green tea extract.

SECONDARY OUTCOMES:
Alanine aminotransferase (ALT) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on ALT.
Aspartate aminotransferase (AST) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on AST.
Total bilirubin (TB) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in liver function based on total bilirubin.
Serum creatinine | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in kidney function based on serum creatinine.
Glomerular filtration rate (GFR) | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in kidney function based on GFR.
Fasting blood glucose | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in blood glucose levels based on fasting blood glucose.
Total cholesterol | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on total cholesterol.
Triglycerides | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on triglycerides.
Low-density lipoprotein (LDL) cholesterol | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on LDL.
High-density lipoprotein (HDL) cholesterol | 0 (baseline; pre-dose), week 2 and week 4 (post-dose)
  To evaluate changes in lipid profile based on HDL.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solnier, Principal Investigator — Isura
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No